CLINICAL TRIAL: NCT06276361
Title: A Single Ascending Dose Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability of a Single Intramuscular Injection of Quarterly Risperidone (QUAR) for Different Formulations and Dose Strengths in Participants With Schizophrenia (QUARTZ Study)
Brief Title: Pharmacokinetics, Safety and Tolerability of Different Formulations and Dose Strengths of Quarterly Risperidone (QUAR) in Patients With Schizophrenia
Acronym: QUARTZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ROV-QUAR-2023-01
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1/2 (Experimental): Patient will recieve oral risperidone for one week followed by a single IM injection of Risperidone QUAR out of two possible formulations (F1/F2) with a level 1 dose.
  Interventions: Drug: Oral risperidone; QUAR F1/2, Dose 1 - Gluteal
- Cohort 1a/2a (Experimental): Patient will recieve oral risperidone for one week followed by a single IM injection of Risperidone QUAR out of two possible formulations (F1/F2) with a level 2 dose.
  Interventions: Drug: Oral risperidone; QUAR F1/2, Dose 2 - Gluteal
- Cohort 1b//2b (Experimental): Patient will recieve oral risperidone for one week followed by a single IM injection of Risperidone QUAR out of two possible formulations (F1/F2) with a level 3 dose.
  Interventions: Drug: Oral risperidone; QUAR F1/2, Dose 3 - Gluteal
- Cohort 1c/2c (Experimental): Patient will recieve oral risperidone for one week followed by a single IM injection of Risperidone QUAR out of two possible formulations (F1/F2) with a level 3 dose.
  Interventions: Drug: Oral risperidone; QUAR F1/2, Dose 3 - Deltoids

INTERVENTIONS:
Drug: Oral risperidone; QUAR F1/2, Dose 1 - Gluteal — Dose level 1
  Arms: Cohort 1/2
Drug: Oral risperidone; QUAR F1/2, Dose 2 - Gluteal — Dose level 2
  Arms: Cohort 1a/2a
Drug: Oral risperidone; QUAR F1/2, Dose 3 - Gluteal — Dose level 3
  Arms: Cohort 1b//2b
Drug: Oral risperidone; QUAR F1/2, Dose 3 - Deltoids — Dose level 3
  Arms: Cohort 1c/2c

SUMMARY:
This is a single ascending dose phase 1 study to evaluate the pharmacokinetics (PK), safety, and tolerability of a single intramuscular (IM) injection of quarterly Risperidone (QUAR) for different formulations and dose strengths in participants with schizophrenia.

DETAILED DESCRIPTION:
The study will assess the PK, safety and tolerability of QUAR when administered as a single IM injection, in patients with schizophrenia. The study will be conducted with 3 different dose strengths and up to two formulations.

After eligibility confirmation, an oral treatment period follow by a washout period will be performed before QUAR IM administration.

The different cohorts will be administered with one of the following dosages of Risperidone QUAR:

Cohort 1/2: Formulation 1 or 2. Dose level 1 (Gluteal); Cohort 1a/2a: Formulation 1 or 2. Dose level 2 (Gluteal); Cohort 1b/2b: Formulation 1 or 2. Dose level 3 (Gluteal); Cohort 1c/2c: Formulation 1 or 2. Dose level 3 (Deltoid);

The progression to the next cohorts will take place after a clinical safety assessment. Several blood samples for plasma pharmacokinetic (PK) assessments will be obtained pre-dose and post-dose. Safety assessments will be conducted at each pre-specified time points.

After assessment of Cohort 1 (formulation 1, Dose Level 1, -gluteus-) progression to the next cohort with same formulation and escalating dose will take place (Cohort 1a -gluteus-). After assessment of Cohort 1a, progression and randomization (gluteus/deltoid) to the next cohorts with same formulation and escalating dose will take place (Cohort 1b -gluteus- and Cohort 1c -deltoid-). In this scenario, none of the Cohorts 2 will be conducted.

If the assessment for Cohort 1 is not adequate, none of the subsequent Cohorts 1 (a/b/c) will be conducted and progression to the next cohort (Cohort 2) with different formulation and same level of dose as Cohort 1 will take place (Cohort 2: Formulation 2, Dose Level 1 -gluteus-). After assessment of Cohort 2, progression to the next cohort with same formulation and escalating dose will take place (Cohort 2a -gluteus-). After assessment of Cohort 2a, progression and randomization (gluteus/deltoid) to the next cohorts with same formulation and escalating dose will take place (Cohort 2b -gluteus- and Cohort 2c -deltoid-).

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent.
* Male or female aged ≥ 18 years to < 65 years with BMI ≥17.0 to ≤35.0 kg/m2
* Current diagnosis of schizophrenia, according to the Diagnostic and DSM-5 criteria.
* Medically stable over the last month, and psychiatrically stable without significant symptom exacerbation over the last three months based on the investigator's judgment
* currently taking oral risperidone as maintenance therapy
* Score of ≤ 4 (moderately ill at most) on the Clinical Global Impression - Severity of Illness (CGI-S)
* If a sexually active female of childbearing potential, using a medically accepted method of birth control.

Exclusion Criteria:

* Presence of an uncontrolled, unstable, clinically significant medical condition that in the opinion of the investigator could interfere with the interpretation of safety and PK evaluations
* If female, a positive serum pregnancy test, or planning to become pregnant between signing informed consent and 1 month after the last dose of study drug or is breastfeeding a child.
* History of neuroleptic malignant syndrome and current or past history of clinically significant tardive dyskinesia.
* The participant has a primary diagnosis other than schizophrenia diagnosis that is primarily responsible for current symptoms and functional impairment
* Positive test result for drugs of abuse or alcohol unless the positive finding can be accounted for by documented prescription use.
* In the investigator's opinion, at imminent risk of committing self-harm or harm to others.
* Unwilling to discontinue any of the prohibited medications prior to the baseline visit or unable to safely washout such medication without significant destabilization or increased risk of self-harm (suicide).
* Receipt study drug in another investigational study in the last 90 days.
* Current participation in any other clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
λz | Following Oral and QUAR administration until day 17 or 196 respectively
  Terminal elimination rate constant
t1/2 | Following Oral and QUAR administration until day 17 or 196 respectively
  Terminal elimination half-life
Tmax | Following Oral and QUAR administration until day 17 or 196 respectively
  Time to peak concentration
Cmax | Following Oral and QUAR administration until day 17 or 196 respectively
  Peak plasma concentration
Cmin | Following Oral and QUAR administration until day 17 or 196 respectively
  Minimum plasma concentration
Clast | Following Oral and QUAR administration until day 17 or 196 respectively
  Last observed plasma concentration
AUC0-t | Following Oral and QUAR administration until day 17 or 196 respectively
  Area under the curve
AUCinf | Following QUAR administration until day 196
  Area under the curve
AUCextrap | Following QUAR administration until day 196
  Area under the curve
Vd/F | Following Oral and QUAR administration until day 17 or 196 respectively
  Apparent volume of distribution
Cl/F | Following Oral and QUAR administration until day 17 or 196 respectively
  Apparent total body clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, Amman, Jordan